CLINICAL TRIAL: NCT05882097
Title: Transform Randomised Control Trial in Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Care Ministries, Philippines (Other)
Responsible Party: Principal Investigator, Lincoln Lau, Director of Research, International Care Ministries, Philippines
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: icmugrct
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Health Behavior; Economic Problems; Values, Social
Keywords: values; livelihood; health; program evaluation; intervention; poverty; poverty reduction; Uganda; randomized control trial
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: This study is a cluster-randomised controlled trial. A total of 4,800 participants from 160 communities will be randomly assigned to one of the two treatment arms: Transform and Control. The treatment will be assigned at the community level, so all participating households in a community will be in the same treatment arm. This will prevent dissemination of information and mixing of control and treatment groups among the participants.
  The RCT will be rolled out in two batches. For each batch (i.e. 40 communities), a list of eligible communities will be drawn up and randomised into one of the treatment arms. To reduce the risk of bias, communities and participants will be recruited before the clusters have been randomly allocated.
Who Masked: Participant
Masking Description: The participants will not know which group they belong to. Due to procedures to implement the study, it is inevitable that the operations team will know who will belong to the control and treatment arms (control participants will not receive the Transform program). This study will be a single masked study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm receiving the Transform program (Experimental): Transform: Participants will receive ICM's Transform program.
  In the treatment arm, the full 15-session Transform program will be delivered once a week for 15 consecutive weeks in a venue located within the community. In each session, there will be 90 minutes lessons on livelihood and health delivered by trained ICM staff. Separately, a voluntary values lesson will be delivered by the host community leader.
  Interventions: Other: Transform program
- Control arm receiving no Transform program (No Intervention): Control: Participants will not receive any intervention during the study period.

INTERVENTIONS:
Other: Transform program — International Care Ministries' (ICM) Transform is a 15-lesson, 15-week long values, health, and livelihood program that targets some of the poorest households in Uganda. The health dimension focuses on increasing health knowledge and behaviours on a range of health topics such as malnutrition, respiratory infection, lifestyle, sanitations, family planning and infant care. The livelihood dimension focuses on increasing the amount and sources of household income. Participants will learn about business ideas and farming techniques to diversify their income sources. Additionally, a savings group will be formed at the end of Transform to promote a sustainable strategy to reduce poverty among the participants. The values dimension will focus on relationships, personal character and decision making aspects of an individual.
  Other Names: Poverty alleviation program
  Arms: Treatment arm receiving the Transform program

SUMMARY:
In recent decades, the poverty rate in Uganda decreased by more than half, from 56% in 1992/1993 to 21.4% in 2019/2020. However, Uganda remains as one of the poorest countries in the world. Recognising that poverty is a multifaceted issue, International Care Ministries (ICM), a non-profit organisation, implements a program called Transform to target households living in poverty from 3 dimensions: values, livelihood and health. ICM first started the Transform program in the Philippines and recently expanded to Uganda and Guatemala. The program includes 15 sessions and delivers them to the participants during the course of a 4-month period. Previously, three randomised control trials found positive impacts of Transform on certain poverty indicators in the Philippines. Although positive impacts were found in the Philippines, the effectiveness of Transform in Uganda is unknown.

DETAILED DESCRIPTION:
International Care Ministries (ICM) is a non-governmental organisation with a mission to reduce the burden of extreme poverty. ICM focused its work in the Philippines for more than 30 years and recently expanded to Uganda and Guatemala. The core poverty alleviation program at ICM is called Transform. Transform focuses on improving values, health and livelihood through a 15-week program (1 lesson per week). ICM has conducted three randomized controlled trials (RCT) in the Philippines. This RCT was designed in response to the expansion of ICM's work in Uganda. Realising the poverty issue that was exacerbated by the COVID-19 pandemic, ICM implemented its first Transform program in Uganda in 2020. As of May 2023, more than 210 communities and 5,921 participants received the Transform program in the regions of Kiboga and Kyankwanzi. Despite the fact that previous RCTs found a positive impact of Transform on certain poverty indicators in the Philippines, the effectiveness of Transform is not known in another context. The Philippines and Uganda are vastly different in terms of their economies, cultures and demographics. This study builds on the previous RCTs and aims to evaluate the Transform program on measures of economic outcomes, social capital, health, hope and spiritual well-being in a different context. Whether there will be similar results in Uganda will deepen perspectives in the universal elements of success that can be further adopted and scaled up in other countries. While a key challenge in poverty alleviation initiatives is the lack of high quality evidence to evaluate the effectiveness of programs, this study will use the gold standard of effectiveness research - RCT, to deepen understanding in the causal impact of the Transform program in another context.

ELIGIBILITY:
Inclusion Criteria:

1. Poverty score of 50 and above in the Philippine Poverty Score Card Survey qualifies the person into Transform. Higher score indicates poorer households.
2. Only the top 30 poorest household will be selected once the community gets approve to host the Transform program.

Exclusion Criteria:

1. Participants who are above the threshold using the poverty score card (less than 50) will be excluded from the study.
2. Households also cannot participate in the study if they have previously received the Transform program, unless the implementation team overrides the score due to specific circumstances that only affect a minority of participants.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in EuroQol-5 Dimension - 5 levels (EQ-5D-5L) at 6 and 12 months | Baseline, 6 and 12 months
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Values are anchored at 1 (full health) and 0 (a state as bad as being dead). Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. Higher value indicate better health state.
Change from baseline in poverty probability index at 6 and 12 months | Baseline, 6 and 12 months
  The Poverty Probability Index (PPI®) is a poverty measurement tool for organizations and businesses with a mission to serve the poor. The answers to 10 questions about a household's characteristics and asset ownership are scored to compute the likelihood ranged from 0 to 1 to indicate how likely the household is living below the poverty line. The higher the probability means that more likely the household is poor.

SECONDARY OUTCOMES:
Change from baseline in duckworth index at 6 and 12 months | Baseline, 6 and 12 months
  Duckworth index measures grit scale on trait-level perseverance and passion for long term goals. This will explore participants characteristic on grit in relations to changes in other variables. The index score ranged from 0 to 5. Higher score indicates greater level of grit.

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln L Lau, PhD, Principal Investigator — University of Toronto
Locations (1):
- ICM Uganda, Kampala, Kibuye, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owori M. Poverty in Uganda: National and regional data and trends. Development Initiatives. https://devinit. org/resources/poverty-uganda-national-and-regional-data-and-trends. 2020 Oct.
- [Background] Bryan G, Choi JJ, Karlan D. Randomizing religion: the impact of Protestant evangelism on economic outcomes. The Quarterly Journal of Economics. 2021 Feb;136(1):293-380.